CLINICAL TRIAL: NCT01551225
Title: Randomized Controlled Trial of Escitalopram Versus Placebo for Patients With Irritable Bowel Syndrome and Panic Disorder
Brief Title: Escitalopram Trial for Irritable Bowel Syndrome (IBS) Patients With Panic Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 102051
Record Dates: First submitted 2011-11-03; First posted 2012-03-12 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-07

CONDITIONS: Irritable Bowel Syndrome; Panic Disorder
Keywords: Randomized controlled trial; Escitalopram; Irritable bowel syndrome; Panic disorder
MeSH Terms: conditions — Irritable Bowel Syndrome; Panic Disorder | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Escitalopram (Active Comparator): 17 or 18 Patients with IBS and panic disorder treated with Escitalopram.
  Interventions: Drug: Escitalopram
- Placebo tablets to Escitalopram (Placebo Comparator): 17 or 18 Patients with IBS and panic disorder treated with placebo.
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Escitalopram — Patients will start at a dosage of 5 mg daily of escitalopram. After the first week of treatment the dosage will be increased to 10 mg daily. During the visits, the dosage can be gradually increased to a maximum of 20 mg daily, depending on the response of the patient.
  Other Names: Lexapro

SUMMARY:
This study will be executed according to a randomized double-blind placebo-controlled trial with two parallel groups, treated over the period of 6 months with escitalopram or placebo.

Hypotheses: Escitalopram is more effective than placebo in the control of gastrointestinal symptoms, in irritable bowel syndrome (IBS) patients with panic disorder. Escitalopram is more effective than placebo in the control of psychiatric symptoms, in IBS patients with panic disorder.

ELIGIBILITY:
Inclusion Criteria:

1. IBS will be diagnosed according to the Rome III criteria by a gastroenterologist.
2. Subtyping of IBS patients will be performed using the following classification according to the Rome III criteria: IBS with constipation (IBS-C), IBS with diarrhea (IBS-D), mixed IBS (IBS-M) or not subtyped IBS (IBS-U).
3. Based on the medical history and previous examination, no other causes for the abdominal complaints can be defined.
4. A panic disorder will be diagnosed based on DSM IV criteria by a psychiatrist.
5. Age above 18 years and under 70 years.
6. Given written informed consent.

Exclusion Criteria:

1. Inability to stop medication that can influence gastrointestinal motility or perception (like loperamide, butylscopolamine, duspatalin, metoclopramide, domperidon, erytromycin), serotonin metabolism (like carbidopa, food supplementation), or epigenetics (like valproic acid), or containing perforated St. John's wort (Hypericum perforatum). In general this medication can be stopped without problems. However, this can increase symptoms. When the increase in symptoms will be to high, this medication will be restarted and the patient excluded form the study.
2. Administration of investigational drugs in the 180 days prior to the study.
3. Major abdominal surgery interfering with gastrointestinal function (uncomplicated appendectomy, cholecystectomy and hysterectomy allowed, and other surgery upon judgement of the principle investigator), epilepsy or (hypo)manic episodes.
4. Pregnancy and lactation.
5. Excessive alcohol consumption (> 20 alcoholic consumptions per week) or drug abuse.
6. Co-intervention or other treatment for IBS or anxiety, with the exception of initial co-intervention with benzodiazepines (alprazolam) contrasting side effects due to SSRI's during the first two weeks of dose elevation.
7. Known prolongation of QT-interval or long-QT-syndrome, other cardiac disease, or use of medication with known prolongation of QT-interval.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal Symptom Rating Scale (GSRS). | Change from baseline in outcome of GSRS at 6 months.
  Gastrointestinal Symptom Rating Scale (GSRS) is a self-assessment questionnaire for gastrointestinal symptoms.
State Trait Anxiety Inventory (STAI). | Change from baseline in outcome of STAI at 6 months.
  State Trait Anxiety Inventory (STAI) is a self-assessment device, which includes separate measures of state and trait anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Kruimel, MD PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands

REFERENCES:
- [Derived] Drukker M, Peters JCH, Vork L, Mujagic Z, Rutten BPF, van Os J, Masclee AAM, Kruimel JW, Leue C. Network approach of mood and functional gastrointestinal symptom dynamics in relation to childhood trauma in patients with irritable bowel syndrome and comorbid panic disorder. J Psychosom Res. 2020 Dec;139:110261. doi: 10.1016/j.jpsychores.2020.110261. Epub 2020 Oct 2. PMID 33038815